CLINICAL TRIAL: NCT06743893
Title: Non Traumatic Chronic Subdural Haematoma in Paediatric Age Groups, Management and Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abo bakr mitwally, principal investigator, Assiut University
Other Study IDs: NTCSDH
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Chronic Non-Traumatic Intracranial Subdural Haemorrhage
Keywords: chronic- subdural haematoma- non traumatic-pediatric age group

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Diagnosis and outcome of non traumatic chronic subdural haematoma in pediatric age groups — Diagnosis and outcome of non traumatic chronic subdural haematoma in pediatric age groups

SUMMARY:
1-Review the management strategies and outcomes in cases of non traumatic chronic subdural haematoma in paediatric age group. 2- Review the underlying causes and risk factors in cases of non traumatic chronic subdural haematoma in paediatric age group

DETAILED DESCRIPTION:
2.4.1- Type of the study: prospective case series study 2.4. 2- Study Setting: Neurosurgery department Assiut university hospital 2.4. 3- Study subjects:

1. Inclusion criteria:

   1-Age less than 18 years. 2-patient with subdural haematoma other than traumatic
2. Exclusion criteria:

   1-Age more than 18 years. 2-patient with traumatic subdural haematoma. 3- patient unfit for surgery

   Patient and method:

   1-General examination. 2- Neurological examination. 3- complete basal investigations. 4-Imaging brain CT scan In paediatric patients with subdural hematoma with an amount of bleeding requiring surgical management, any underlying comorbidities should be investigated regardless of the presence of a history of trauma. While investigating systemic diseases, special attention should be paid to the presence of arachnoid cysts or disruption in cerebrospinal fluid dynamics along with a history of hematologic diseases Data on patient sex, age, bleeding location, type of hematoma based on computed tomography imaging, surgical treatment, presenting symptoms, presence of comorbidities, Glasgow Coma Scale, platelets counts, and international normalized ratio values were recorded There will be file to collect data ( patient data sheet)of the patient: involving personal data and detailed history and detailed general and neurological examinations and all general investigations and specific according to her underlying medical disorders ( risk factor and cause of non traumatic subdural haematoma) and type of treatment that received and report of ct scan and mri Symptoms of subdural haematoma: Drowsy/unconscious , Poor feeding , Irritability , Fits , Pallor , Floppiness , Vomiting , Sudden collapse, Breathing difficulties , Large head , Apnoea , Delayed development Neurological assessment plus Glasgow Coma Scale(paediatric GCS and pupillary reactivity) Investigations: CT scan brain MRI BRAIN : cranial subdural haematoma site and location , size in cm, detected midline shift ,uni or bilateral subdural haematoma, haematoma density , haematoma thickness plus other cranial bleeding or pathology or other spinal cord bleeding or pathology All blood investigations including cbc , coagulation profile , liver ,renal functions , all investigations related to underlying medical or neurological or neurosurgical disorder.

   Treatment: admission either in intensive care unit ,or in the department and type of treatment either medical with conservative involving dexamethasone plus or minus atrovostatins(2.5-5 mg atorvastatin daily combined with dexamethasone with stepwise-decreasing dosing for a total of 4 weeks) Or surgical in the form of burr hole trepanation (Burr-hole drainage (BHD), craniectomy and craniotomy After treatment follow up for 2 days , one month and three months post operative.
3. Sample Size Calculation: 30 cases according previous case series studies in these rare disease and according to sample size calculation.

2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):CT scan brain MRI BRAIN detected site and location of cranial subdural haematoma ,midline shift uni or bilateral subdural haematoma, haematoma density , haematoma thickness plus other cranial bleeding or pathology or other spinal cord bleeding or pathology All blood investigations including cbc , coagulation profile , liver ,renal functions , all investigations related to underlying medical or neurological or neurosurgical disorder There will be file to collect data ( patient data sheet)of the patient involving personal data and detailed history and detailed general and neurological examinations and all general investigations and specific according to her underlying medical disorders ( risk factor and cause of non traumatic cranial subdural haematoma) and type of treatment that received and report of ct scan and mri

ELIGIBILITY:
Inclusion Criteria:1-Age less than 18 years. 2-patient with subdural haematoma other than traumatic -

Exclusion Criteria:1-Age more than 18 years. 2-patient with traumatic subdural haematoma. 3- patient unfit for surgery

-

Ages: 1 Hour to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric age group from first hour after birth of newborn till 18 years old
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
diagnosis and outcome of different types of treatment of non traumatic chronic subdural haematoma in paediatric age group in within one year. | one year
  diagnosis and outcome of different types of treatment of non traumatic chronic subdural haematoma in paediatric age group.

SECONDARY OUTCOMES:
Secondary (subsidiary): the underlying risk factors and possible relation to non traumatic chronic subdural haematoma in paediatric age group and how to decrease its recurrence | one year
  Secondary (subsidiary): the underlying risk factors and possible relation to non traumatic chronic subdural haematoma in paediatric age group and how to decrease its recurrence

IPD SHARING:
Plan to Share IPD: Undecided